CLINICAL TRIAL: NCT01785732
Title: Renal Sympathetic Denervation and Insulin Sensitivity (RENSYMPIS Study)
Acronym: RENSYMPIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SA-007
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal denervation (Active Comparator): Patients are randomized to renal denervation
  Interventions: Procedure: Renal Denervation
- Optimization of medical therapy (No Intervention): Antihypertensive treatment is optimized

INTERVENTIONS:
Procedure: Renal Denervation — Sympathetic renal denervation via renal arteries
  Arms: Renal denervation

SUMMARY:
Hypertension is a major risk factor for stroke and cardiovascular mortality. Catheter- based renal denervation causes substantial and sustained blood- pressure reduction in patients with resistant hypertension.

The purpose of RENSYMPIS is to study the effects of renal denervation on:

1. Cardiovascular function
2. Metabolic factors
3. Inflammatory and endocrine factors
4. Coagulation
5. Sleep

ELIGIBILITY:
Inclusion Criteria:

* Resistant Hypertension (systolic blood pressure >160mmHg and 3 or more antihypertensive agents in use)
* Age 30- 69 years
* Written informed consent

Exclusion Criteria:

* Secondary hypertension
* Pseudohypertension
* Pregnancy
* Renal insufficiency (GFR <45ml/min)
* Clinically significant stenotic valvular disease
* Oral anticoagulation
* CCS III-IV symptoms or CABG/PCI in previous 6 months
* Prior stroke
* Contrast agent allergy
* inappropriate renal artery anatomy (< 4mm diameter, < 20mm length)

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Office blood pressure | 2 years

SECONDARY OUTCOMES:
Ambulatory blood pressure | 2 years
Insulin resistance | 2 years
Endothelial function | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Satakunta Central Hospital, Pori, Finland